CLINICAL TRIAL: NCT07232173
Title: Comparative Study Between Pericapsular Nerve Group Block (PENG) Versus Suprainguinal Fascia Iliaca Compartment Block (SFIC) in Perioperative Hip Surgery
Brief Title: Comparative Study Between Pericapsular Nerve Group Block (PENG) Versus Suprainguinal Fascia Iliaca Compartment Block (SIFIC) in Perioperative Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Noser, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU M D 235/2020
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Anesthesia; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound-guided pericapsular nerve group block PENG (Active Comparator)
  Interventions: Procedure: Pericapsular Nerve Group Block (PENG)
- ultrasound-guided supra-inguinal fascia iliaca block SFIC (Active Comparator)
  Interventions: Procedure: Suprainguinal Fascia Iliaca compartment Block (SIFIC)

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block (PENG) — Participants in the PENG group first received their study medication, administered over a 1-minute interval, 5 minutes prior to the initiation of spinal anesthesia. For the block itself, an in-plane ultrasound-guided approach was utilized. Following the creation of a skin wheal, an echogenic, 10-centimeter, 21-gauge needle was carefully advanced in a lateral-to-medial trajectory. The local anesthetic, 20 mL of .5% ropivacaine, was then accurately injected into the fascial plane located anterior to the psoas tendon and posterior to the pubic ramus.
  Arms: ultrasound-guided pericapsular nerve group block PENG
Procedure: Suprainguinal Fascia Iliaca compartment Block (SIFIC) — The SFIC group block began with a skin wheal and employed an in-plane needle insertion. Once the needle successfully pierced the fascia iliaca, a small 2 mL volume of saline was initially injected. This served as a hydraulic confirmation of the correct needle tip placement within the compartment.
  Arms: ultrasound-guided supra-inguinal fascia iliaca block SFIC

SUMMARY:
The hip joint is the largest and one of the most stable joints in the human body. It bears the majority of the body's weight during both dynamic and static activities, making it highly susceptible to degenerative diseases, particularly in the elderly population. In advanced cases, total hip arthroplasty (THA) is often required-currently ranking as the second most common joint replacement procedure worldwide.

Despite its clinical success, it is estimated that 7-28% of patients experience chronic postoperative pain following THA. This persistent pain significantly impairs quality of life and is receiving growing attention from healthcare professionals. Evidence suggests that unmanaged acute surgical pain is a major risk factor for the development of chronic postoperative pain, underscoring the importance of effective perioperative analgesia. Given the adverse effects associated with opioids, regional anesthesia techniques are increasingly favored for pain management.

Among these, the fascia iliaca compartment block (FICB) has been widely used to reduce postoperative pain intensity, although it carries potential drawbacks such as motor weakness or a need for supplemental opioid use. Recent anatomical studies by Short et al. have identified the anterior capsule of the hip joint as being innervated by the pericapsular nerve group (PNG) including the obturator nerve, accessory obturator nerve, and femoral nerve. The anatomical accessibility of these nerves has enabled the development of the pericapsular nerve group (PENG) block, a motor-sparing regional anesthesia technique that offers targeted analgesia by delivering local anesthetics into the myofascial plane between the psoas muscle and the superior pubic ramus.

While both FICB and PENG blocks are widely used in total hip replacement surgeries, comparative evidence evaluating their efficacy remains limited. Therefore, this study aims to compare the analgesic effectiveness of FICB and PENG blocks during the preoperative and postoperative phases of total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* non-pathologic hip fractures
* underwent total hip arthroplasty (THA) or hemiarthroplasty at Ain Shams University Hospitals
* physical status I, II and III according to the American Society of Anesthesiologists (ASA) classification.

Exclusion Criteria:

* pathological fracture
* allergy to study drugs.
* ASA IV (a patient with severe systemic disease that is a constant threat to life)
* bleeding tendencies
* dementia or any mental disability
* having sepsis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
onset of analgesia | Assessed before the block and every 3 minutes from blocking for 30 minutes afterwards.
  defined as an NRS of 3 or less at rest and during passive 20° limb elevation.

SECONDARY OUTCOMES:
NRS over 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided